CLINICAL TRIAL: NCT02660164
Title: A Study to Assess the Effectiveness of the Nautilus BrainPulse™ as an Aid in the Diagnosis of Concussion
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JMC-1501
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Concussion
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: High-Risk of Concussion: Middle school, high school and college athletes of either gender participating in sports where high-risk of concussion is anticipated: football, soccer, lacrosse, hockey, basketball, ice hockey, field hockey, rugby, cheerleading, boxing, and gymnastics.
  Interventions: Device: Nautilus BrainPulse Recording
- Cohort B: Low-Risk of Concussion: Middle school, high school and college athletes of either gender participating in sports where low-risk of concussion is anticipated: swimming, track, volleyball, baseball, softball and golf.
  Interventions: Device: Nautilus BrainPulse Recording

INTERVENTIONS:
Device: Nautilus BrainPulse Recording — Comparison of Nautilus BrainPulse recordings in subjects who have a concussive event (Cohort A) to Nautilus BrainPulse recording in subjects who do not experience a concussive events (Cohort B or matched subjects to Cohort A). Recordings are obtained over a 2 week period every 2 to 3 days (at least 5 recordings per subject).

SUMMARY:
The objective of the study is to evaluate, in a blinded fashion, the effectiveness of the Nautilus BrainPulse device when used as an aid in the diagnosis of concussion.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, blinded, matched control study of young athletes (ages 10-25 years old) in competitive sports (Cohort A: higher-risk of concussion, Cohort B: lower-risk of concussion) to assess the effectiveness of the Nautilus BrainPulse device when used as an aid in the diagnosis of concussion.

The Nautilus BrainPulse is intended for use on a patient's head to non-invasively detect, amplify and capture the brain pulse, the brain motion caused by pulsatile blood flow from the cardiac cycle. The Nautilus BrainPulse analyzes the captured data to provide an aid in diagnosing an episode of concussion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 10 and 25 years of age (middle school, high school or college-age)
2. Team member, where the team meets at least twice a week
3. Willing and able to participate in all study evaluations and allow access to medical testing and records
4. Signed informed consent, or have a legally authorized representative willing to provide informed consent on behalf of the subject if the subject is a minor

Exclusion Criteria:

1. Documented history of a concussion diagnosed by a physician in the last two months assessed via interview with athlete
2. Known history of any cognitive deficits that diminish ability to administer study assessments, such as SCAT3™
3. Wound on the head in the area of one of the Nautilus BrainPulse sensors that would impede use of the Nautilus BrainPulse device
4. Inability to obtain a valid SCAT3 and ImPACT® baseline assessment of concussion
5. Any serious medical, social or psychological condition that in the opinion of the investigator would impair ability to provide informed consent or otherwise disqualify a patient from participation

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cohort A: High-Risk of Concussion Middle school, high school and college athletes of either gender participating in sports where high-risk of concussion is anticipated: football, soccer, lacrosse, hockey, basketball, ice hockey, field hockey, rugby, cheerleading, boxing, and gymnastics.
  Cohort B: Low-Risk of Concussion Middle school, high school and college athletes of either gender participating in sports where low-risk of concussion is anticipated: swimming, track, volleyball, baseball, softball and golf.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Nautilus Brain Pulse in detecting concussion as compared to adjudication by a panel of medical experts | 10 days
  Sensitivity and Specificity of the Nautilus BrainPulse in detecting the number of subjects experiencing concussion as compared to the number of subjects with concussion as adjudicated by a panel of medical experts. BrainPulse measurement data will be aggregated by subject over the first 10-days of recording after the concussive event, or for subjects in the Control arm, after their selection as a control subject.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Abrams, MD,, Principal Investigator — University of California San Francisco Medical Center
Locations (4):
- United States (4):
  - Meli Orthopedic Centers of Excellence, Fort Lauderdale, Florida
  - Community Hospital, Munster, Indiana
  - Louisiana State University, Baton Rouge, Louisiana
  - University of Wyoming, Laramie, Wyoming